CLINICAL TRIAL: NCT06166043
Title: Evaluation of the Efficiency of the Nurse Follow-up Program Supported With Web Based Education in Managing Fatigue in Patient With Multiple Sclerosis
Brief Title: The Effect of the Nurses Support Program on Fatigue in MS Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, GİZEM YAĞMUR YALÇIN, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/13
Record Dates: First submitted 2023-08-24; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis; Fatigue; Sleep Hygiene; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: Patients will receive standard care first. The same group of patients will later be included in the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NURSE FOLLOW-UP PROGRAM SUPPORTED WITH WEB-BASED EDUCATION IN (Experimental): An online training consisting of 10 sessions in total for 5 weeks will be given to the patients in order to improve their fatigue management skills. In addition to this training, they will receive a nurse support program.
  Interventions: Behavioral: NURSE FOLLOW-UP PROGRAM SUPPORTED WITH WEB-BASED EDUCATION

INTERVENTIONS:
Behavioral: NURSE FOLLOW-UP PROGRAM SUPPORTED WITH WEB-BASED EDUCATION — An online training consisting of 10 sessions in total for 5 weeks will be given to the patients in order to improve their fatigue management skills. In addition to this training, they will receive a nurse support program.

SUMMARY:
The research will be carried out as a randomized controlled experimental study to examine the effect of a nursing support program supported by a Web-based education program on the management of fatigue symptoms of patients who are under treatment and care in the Multiple Sclerosis clinic of a university hospital.Patients will receive 5 weeks of standard care. At the end of 5 weeks, they will enter a training program. After this online training program, which will be 5 weeks and 2 sessions per week, the change in the patients' fatigue, sleep quality and quality of life will be analyzed.

DETAILED DESCRIPTION:
Interventions

Groups will be determined in accordance with the randomisation method within the scope of the research for patients who voluntarily agree to participate in the research and meet the inclusion criteria. After the patient is informed about the research in accordance with the group selected, both verbal and written consent will be obtained through the "Voluntary Consent Form".

Control Group: The selected patients will first be included in the control group. Patients will be measured before the study and will receive standard care for 5 weeks without any intervention. At the end of 5 weeks, the measurements of the patients will be repeated. Patients will then be included in the case group. Fatigue Severity Scale, Pittsburg Sleep Quality Scale, EQ5D Quality of Life Scale will be applied to the patients at the beginning and after 5 weeks of receiving standard care.

Case Group: The case group will be included in a 5-week programme including a web-based training programme and nurse follow-up system. This training package, which is determined as 2 days a week for 5 weeks and each session will last 50 minutes, will be carried out through the zoom programme because it is easy to use and adapt. The content of the training is based on fatigue management, taking into account the relevant factors in parallel with the literature. Before the training starts, the patients will be fitted with a smart watch and their step counts and sleep patterns (sleep time, what time they go to bed, deep sleep and light sleep hours) will be monitored for 7 days and this information will be obtained from the patient on a daily basis. They will be informed that they should never take the watch off their wrists and make sure that it works in a healthy way. At the same time, the watch of the researcher and the watch of the participants will be matched to make sure that the watches of the patients are working and measuring simultaneously. Fatigue Severity Scale, Pittsburg Sleep Quality Scale, EQ5D Quality of Life Scale will be applied to the patients. In order to see the behavioural change more clearly after the end of the training, the clock measurements of the patients will be recorded again for 7 days after 1 month and the specified scales will be applied again. At 3 and 6 months, only the scales will be applied again.

Web-based Education Programme After the interviews with the patients, a day and time suitable for the patients will be determined.

WEEK 1: Starting the session, summarising the education plan to be made to the patients, learning the expectations of the patients from the education and ensuring the interaction of mutual group participants. The definition of Multiple Sclerosis, the causes of fatigue in MS and the definition of fatigue will be explained with a Powerpoint presentation (ppt) prepared with literature information. Then patients will be given time to share their experiences. Participants' questions will be answered.

WEEK 2: Training on sleep hygiene and physical exercise will be given. In the first training session of the week, sleep hygiene will be explained. In the second session, exercise will be performed simultaneously with the patients. An exercise plan consisting of stretching-resistance-tension-balance sets will be applied. Patients will be advised to walk for 25 minutes 3 days a week for exercise and the implementation status will be provided and monitored simultaneously with smart watch data.

WEEK 3: Energy conservation training will be explained to patients using interactive methods in the form of Ppt. (Patients will be able to answer the questions asked simultaneously using their mobile phones and patient participation will be ensured by making it visible on the screen by all users) Energy conservation training; It was developed by Packer and colleagues for individuals with chronic diseases that cause fatigue (Blikman et al., 2017). This training includes strategies such as the importance of rest, storing and using energy, appropriate use of body mechanics, organising activities, using assistive technology, setting priorities and standards, and maintaining balance in daily life. It aims to ensure that the individual uses the available energy at the optimum level while fulfilling the activities in daily life.

WEEK 4: Time Management training will be given. It aims to ensure that the individual uses his/her current energy at the optimum level by determining planned and priorities while performing activities in daily life (Audulv et al., 2021).

WEEK 5: Previous trainings will be summarised, patients' feedback will be received. If they have questions, they will be answered. The training will be terminated by ensuring interaction between patients.

Nurse Support Programme

Patients will be called twice a week using a practice list prepared by the researcher and it will be monitored whether the activities on this list are implemented or not. Patients will be reminded of the training time and day by sending SMS 1 day before and 1 hour before the training time, and patients will be prevented from overlooking this information thanks to the simultaneous notification to the smart watch they use. In the same process, patients will be able to reach their nurses via SMS or call at any time with the mobile phone number provided. This support package also includes the follow-up of patients' medication, paperwork on the hospital side, follow-up of patients' appointment processes, follow-up of blood tests during medication use and ensuring that the results are evaluated by appropriate people. Guidance and motivational support will be provided to patients in their processes within the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MS according to McDonald diagnostic criteria at least 6 months ago Being over 18 years old Having voluntarily agreed to participate in the study Having a score below 18 points from the depression tests (Beck Depression Scale), EDSS score <5

Exclusion Criteria:

* Presence of a diagnosed psychological illness Having had an attack in the last 3 months Having a score below 24 points in the Mini Mental test evaluation The patient's heart failure Having thyroid hormone imbalance Having uncontrolled and unfollowed anemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Fatigue levels | The first measurements are made on the patients included in the study. After 5 weeks, the same measurements are made again. The same measurements are made for the patients included in the training 9 weeks and 17 weeks after the start of the training.
  Fatigue levels of the patients will be measured before and after the education.Patients' fatigue levels will be measured using the fatigue severity scale. The scale consists of 9 items. It is a scale that the patient can fill in themself.

SECONDARY OUTCOMES:
sleep quality levels | The first measurements are made on the patients included in the study. After 5 weeks, the same measurements are made again. The same measurements are made for the patients included in the training 9 weeks and 17 weeks after the start of the training.
  The sleep quality of the patients will be evaluated with the Pittsburg sleep quality scale, which is a 24-item scale in total. Each item in the scale is scored between 0-3 and the total score varies between 0-21. A total PDQI score greater than five indicates that the sleep quality of the individual is inadequate.
quality of life levels | The first measurements are made on the patients included in the study. After 5 weeks, the same measurements are made again. The same measurements are made for the patients included in the training 9 weeks and 17 weeks after the start of the training.
  The EQ-5D quality of life scale will be used to measure quality of life. The EQ-5D was developed by the EuroQol Group, an international, interdisciplinary group established in 1987 to investigate issues related to the assessment of health. It has been translated into more than 60 languages and is used worldwide. The reliability and validity of the EQ-5D has been established both in general (Brooks & De Charro, 1996) and in disease-specific groups (Öster et al., 2009; Schrag et al., 2000; Schweikert et al., 2006).
  The EQ-5D descriptive system includes five questions covering five dimensions: mobility, self-care, usual activities, pain and anxiety/depression. For each dimension, participants rate their health by reporting whether they experience 1 = "none", 2 = "moderate" or 3 = "extreme problems".Participants receive a score between 0.59 and 1. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Gizem Yağmur Yalçın, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yalcin GY, Tulek Z, Kurtuncu M. Effect of a nurse-led online patient support program on fatigue, sleep and quality of life in patients with multiple sclerosis: a quasi-experimental study. BMC Neurol. 2025 May 31;25(1):238. doi: 10.1186/s12883-025-04248-8. PMID 40450247